CLINICAL TRIAL: NCT01166854
Title: Characterization of Familial Myopathy and Paget Disease of Bone
Status: Recruiting | Type: Observational
Sponsor: University of California, Irvine (Other)
Collaborators: Beckman Laser Institute University of California Irvine (Other)
Responsible Party: Principal Investigator, Virginia Kimonis, Virginia Kimonis, MD, MRCP, University of California, Irvine
Other Study IDs: 20075832
Record Dates: First submitted 2010-07-20; First posted 2010-07-21 (Estimated); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Muscle Disorder; Bone Disorder
Keywords: muscle and bone disease
MeSH Terms: conditions — Muscular Diseases; Bone Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Muscle weakness: Diffuse Optical Spectroscopy
  Interventions: Device: Diffuse Optical Spectroscopy

INTERVENTIONS:
Device: Diffuse Optical Spectroscopy — Diffuse Optical Spectroscopy

SUMMARY:
The researcher wants to explore the genetic causes of muscle disease. The researcher is particularly interested in muscle disorders that occur in combination with diseases of bone that appear to be passed on from generation to generation.

Diffuse Optical Spectroscopy will measure the concentrations of blood, water, and lipids (fats, for example) in your tissues. This device essentially measures the color of tissues in order to determine tissue physiology (its physical and chemical processes).

DETAILED DESCRIPTION:
Diffuse Optical Spectroscopy, the technique is fast and painless and was developed at the University of California, Irvine. The Diffuse Optical Spectroscopy instrument is actively involved in research studies, but is not yet a part of routine clinical practice. The result of this study will aid similar research projects that seek to improve our understanding of how tissues work and how alterations in metabolism affect long-term health.

TheDiffuse Optical Spectroscopy measurement consists of placing a probe onto the surface of your body (calf, bicep, or head). This probe will be secured by either gentle hand pressure or fastened to your skin using clinically-approved wraps such as Coban/wrap bandages or medical adhesive tape and medical glues. Several dots will be made on your skin outlining the probe with a surgical felt tip marker. This is so we would be able to put the probe again on the same spot in case we needed to interrupt the measurement. The probe looks like a bar code scanner in a supermarket and it shines infrared light on your skin. There is no radiation involved with this light. In some cases where light signals are low, the optical detector will be placed directly onto your skin (but contained within an electronically shielded casing, and placed inside another plastic casing). (not offered during pregnancy).

ELIGIBILITY:
Inclusion Criteria: Male or Female age 18 and older

* diagnose of Muscle or bone disorders
* with a combination of medical problems including muscle and bone disease and their family members.

Exclusion Criteria:

* under 18 year of age
* unrelated diagnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study Population will be selected from Dr. Kimonis outpatient clinic at University of California Irvine.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2010-06-18 (Actual); Primary Completion 2030-06 (Estimated); Study Completion 2030-06 (Estimated)

PRIMARY OUTCOMES:
muscle disease | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Virginia Kimonis, MD, Principal Investigator — Beckman Laser Institute University of California Irvine; Bruce Tromberg, PhD, Study Director — Beckman Laser Institute University of California Irvine
Locations (1):
- Hewitt Hall, Irvine, California, United States